CLINICAL TRIAL: NCT02078765
Title: Nocturnal Blood Pressure in Hypertension, Obstructive Sleep Apnea and Healthy Subjects - Central and Peripheral 24-h Blood Pressure
Brief Title: Nocturnal Blood Pressure and Hypertension - Central and Peripheral 24-h Blood Pressure.
Acronym: HOSA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, professor, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Other Study IDs: BGH-2-2013; M-2013-303-13 (Other: The Regional Committee of health Reseach Ethics)
Record Dates: First submitted 2014-03-01; First posted 2014-03-05 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension; Chronic Kidneys Disease; Obstructive Sleep Apnea
Keywords: hypertension; chronic kidneys disease; obstructive sleep apnea; 24-h blood pressure; central blood pressure; peripheral blood pressure
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood, serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hypertension: 75 patients with hypertension and chronic kidney disease (CKD stage I-II)
- healthy subjects: 75 healthy subjects

SUMMARY:
A new study have shown that high night time blood pressure (BP) and/or non-dipping (lack of fall in BP during night time) is a strong predictor for the risk of cardiovascular disease and mortality in patients with hypertension. Three factors seem to affect the night time BP: chronic kidney disease, obstructive sleep apnea (OSA) and the way ambulatory blood pressure is monitored.

Hypothesis:

Central 24-h blood pressure monitoring is a better way of monitoring blood pressure than conventional peripheral monitoring.

In hypertension, chronic kidney disease and obstructive sleep apnea (OSA) the night time blood pressure is elevated, and is OSA the elevation is correlated to the severity of OSA.

In OSA the kidneys handling of salt and water is disturbed. In OSA there is disturbances in hormonal balance.

DETAILED DESCRIPTION:
75 patients with hypertension and chronic kidney disease (CKD I-II) and 75 healthy subjects is examined with both central and peripheral 24 hours blood pressure monitoring, 1 night home polygraphy to determine whether the subject has obstructive sleep apnea (OSA), and if so the degree (apnea hypopnea index, AHI), blood and urine samples to determine levels of urine aquaporine2 (u-AQP2), urine endothelial sodium channel (u-EnaC), plasma renin concentration (PRC), plasma angiotensin II (p-AngII), plasma aldosterone (p-aldosterone), plasma vasopressin (p-AVP) and plasma endothelin (p-endothelin).

Hypothesis:

Central 24-h BP monitoring provides another measure of daily fluctuations in blood pressure than peripheral 24-h BP monitoring, because this measurement is painless and does not interfere with activities in the daytime or night-time sleep.

In hypertension, chronic kidney disease and OSA the decease in nocturnal BP is lower than i healthy subjects.

In OSA the decrease in the nocturnal BP is inversely correlated with the severity of OSA.

In OSA is the renal tubular absorption of water and sodium abnormal with increased tubular absorption of water with AQP2 and of sodium by ENAC.

In OSA, there is increased activity of the renin-angiotensin-aldosterone system, increased endothelin in plasma and increased vasopressin in plasma.

ELIGIBILITY:
Group 1:

Inclusion Criteria:

* Chronic kidney disease (CKD stage I and II), estimated glomerule filtration rate (eGFR) 60-90 ml/min/1.73 m2 or eGFR> 90 ml/min/1.73 m2 and proteinuria or other signs of kidney damage.
* Hypertension (BP by ambulatory or home blood pressure> 135/85 mmHg, or consultation blood pressure> 140/90 mmHg).
* Both men and women
* 55-70 years
* A completed consent form

Exclusion Criteria:

* Lack of desire to participate
* In the treatment of OSA
* Malignant disease
* Abuse of drugs or alcohol
* Pregnant and breastfeeding
* Incompensated heart failure
* Atrial fibrillation
* Liver disease (Alanine aminotransferase (ALT)> 200)
* Severe chronic obstructive pulmonary disease (COPD) (Forced expiratory volume in 1 second <50% predicted)
* eGFR <60 ml/min/1.73 m2
* Blood pressure difference between the right and left arm> 10/10 mmHg

Group 2 - Healthy subjects

Inclusion Criteria:

* Healthy subjects men and women
* age 55 - 70 years
* Body mass index within the normal range, between 18.5 to 25.0 kg/m2

Exclusion Criteria:

* Arterial hypertension, ambulatory blood pressure> 130 mmHg systolic and / or 80 mmHg diastolic.

  * a history or clinical signs of cardial, pulmonary, hepato, renal, endocrine, cerebral or neoplastic disorders
  * Alcohol abuse, ie. > 14 drinks / week for women and> 21/uge for men
  * Substance abuse
  * Medical treatment apart from oral contraceptives
  * Smoking
  * Pregnancy or breastfeeding
  * Lack of desire to participate
  * Clinically significant, discrepant results of blood or urine sample at inclusion study (B-hemoglobin and B-White blood cell count, p-sodium, p-potassium, p-creatinine, p-ALT, p-bilirubin , p-Alkaline phosphatase, p-cholesterol, p-albumin or b-glucose and urine for hematuria, albuminuria or glucosuria)
  * Clinically significant variations in the electrocardiogram
  * Blood Donation for the past month preceding the day on the first attempt sequence
  * Blood pressure difference between the right and left arm> 10/10 mmHg.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: 75 patients with hypertension, recruited from another study in the Holstebro Area, contacted by letter.
  Group 2: healthy subjects are recruited though posters in public and private companies as well as advertising in local media.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
decrease in central systolic blood pressure at night | < 24 hours
  The difference in the decrease in systolic BP at night by peripheral 24-h BP between patients with hypertension and healthy subjects.

SECONDARY OUTCOMES:
decrease in central systolic blood pressure at night | < 24 hours
  The difference in the decrease in systolic BP at night by the central 24-h BP between patients with hypertension and healthy subjects.
difference i blood pressure levels throughout the day | < 24 hours
  The difference in systolic blood pressure and diastolic blood pressure throughout the day, in the daytime and in nighttime between peripheral 24-h and central 24-h monitoring in both patients and healthy.
The correlation between the decrease in nighttime BP on one side and severity of OSA and BP in the daytime on the other. | < 24 hours
  The correlation between the decrease in nighttime BP on one side and severity of OSA and BP in the daytime on the other.
u-AQP2 and u-ENac | 24 hours
  In 24-h urine samples
PRC, p-AngII, p-aldosterone, p-AVP, p-endothelin | < 1 hour
  blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Research and Medicine, Holstebro Regional Hospital, Holstebro, Holstebro, Denmark